CLINICAL TRIAL: NCT02351258
Title: Community Central Line Infection Prevention Trial
Acronym: CCLIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB00046284; R01HS022870 (AHRQ)
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Results first posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Infection
Keywords: Pediatrics; Medical Oncology; Catheters; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care only, then Usual Care + 70% Isopropyl Alcohol (Experimental): Usual care for central line while patients are at home and then switch to usual care plus 70% isopropyl alcohol after washout.
  Interventions: Device: 70% Isopropyl alcohol embedded caps; Other: Usual Care
- Usual Care + 70% Isopropyl Alcohol, then Usual Care only (Experimental): Use of 70% isopropyl alcohol embedded caps on central lines in addition to usual care of central line in the home setting and then switch to usual care only after washout.
  Interventions: Device: 70% Isopropyl alcohol embedded caps; Other: Usual Care

INTERVENTIONS:
Device: 70% Isopropyl alcohol embedded caps — Protective cap on central lines
  Other Names: Curos Cap by Ivera Medical Corporation
Other: Usual Care — This involves the Best Practice Central Line Maintenance Care Bundle which includes;
  1. Daily assessment whether central line is needed
  2. Central line Site Care
  3. Central line Hub/Cap/Tubing Care

SUMMARY:
The overall goal of this Community Central Line Infection Prevention (CCLIP) trial, supported by grant R01 HS022870 from the Agency for Healthcare Research and Quality, is to determine whether use of a promising new intervention, namely 70% isopropyl alcohol embedded protective caps on central lines, in the home setting is associated with a reduction in ambulatory central line-associated bloodstream infections (CLABSI) in a high-risk population of pediatric hematology/oncology patients. Despite successes in CLABSI reduction efforts for inpatients, it remains unknown what generalizable best practices should be with chronic central lines in the home setting and how effective involving patients and caregivers across multiple institutions in CLABSI reduction efforts will be. This research will involve a cluster-randomized, cross-over design, clinical trial. This proposal will focus on the caregivers integral to ambulatory pediatric central line care: patients and families. The specific aims of the proposed research program are:

Specific Aim #1: Evaluate whether use of 70% isopropyl alcohol embedded protective caps on central lines reduces the rate of CLABSI in ambulatory pediatric hematology/oncology patients.

Hypothesis: Use of 70% isopropyl alcohol embedded protective caps on central lines will be associated with at least a 25% reduction in the ambulatory CLABSI rate for pediatric hematology/oncology patients.

Specific Aim #2: Evaluate whether use of 70% isopropyl alcohol embedded protective caps on central lines reduces the rate of all positive blood cultures in ambulatory pediatric hematology/oncology patients.

Hypothesis: Use of 70% isopropyl alcohol embedded protective caps on central lines will be associated with at least a 25% reduction in the positive blood culture rate at home for pediatric hematology/oncology patients.

Specific Aim #3: Evaluate whether the use of 70% isopropyl alcohol embedded protective caps on central lines changes the distribution of bacteria isolated from blood cultures of pediatric hematology/oncology patients.

Hypothesis: Use of 70% isopropyl alcohol embedded protective caps on central lines will reduce Gram-positive CLABSI, secondary blood steam infections, and single positive blood cultures at home for pediatric hematology/oncology patients.

DETAILED DESCRIPTION:
Study Design and Population: The proposed study will use a cluster-randomized, 2 period crossover design, clinical trial to evaluate a promising new intervention, namely 70% isopropyl alcohol embedded protective caps, to reduce CLABSIs, 2ndry BSI, and SPBC at home for chronic central lines in pediatric hematology/oncology patients. The Control Arm will involve "usual care" for ambulatory central lines per institutional policy and the Intervention Arm will add use of 70% isopropyl alcohol embedded protective caps to "usual care. Each participating institution will be randomly assigned to either the intervention or control phase of the design for the first 12 months of the study. There will then be a 3 month wash out period, followed by each institution then implementing either the control or intervention phase for another 12 months such that each institution will complete 12 months each in the intervention arm and the control arms of the study.

Sixteen pediatric hematology/oncology institutions will serve as the core population for this proposal and unit of randomization. All ambulatory patients taken care of by these pediatric hematology/oncology clinics at these institutions will be eligible for this study. The only inclusion criteria will be presence of an external central line. Given the intervention is a protective cap for central line access ports, patients who only have a totally implanted port as their central venous access will not be eligible for this study as the intervention is not physically applicable to such central lines.

The intervention the investigators will deploy is the CUROS® brand of 70% isopropyl alcohol embedded protective caps for central lines. These caps are manufactured by Ivera Medical Corporation. As in kind contribution to this proposed study, Ivera Medical Corporation has agreed to donate and distribute all needed CUROS® caps to the participating institutions for the duration of this study. If any of the participating teams wishes to instead use a comparable brand of 70% isopropyl alcohol embedded protective caps for central lines that will be permitted.

Distribution of the CUROS® caps will be accomplished within the clinics of each participating institution and compliance with the intervention at homes will be monitored by clinic staff via tracking counts of CUROS® caps dispensed to families. Children with chronic hematologic/oncologic conditions are seen frequently in clinic, often up to every week. Clinic staff can distribute and track volume of CUROS® caps dispensed to each family/patient, with the family/patient can report back each visit on the volume of CUROS® caps utilized. This will ensure reliable distribution to the families/patients, provide a face to face educational opportunity to ensure proper application of the CUROS® cap, and provide compliance opportunities via counts of CUROS® caps utilized.

This proposal will involve a cluster-randomized, 2 period crossover design, clinical trial. Given this proposal's focus on reducing central line infections at home, the main facilitators of best practice use of these caps at home will be the families and patients themselves. The research team will spread the needed additional education, tools, data, analyses, and support for this proposal.

Study Organization and Timeline: The work will build on the partnership between the pediatric quality improvement research group at Johns Hopkins University and the vendor Ivera Medical Corporation, maker of the CUROS® brand 70% isopropyl alcohol embedded protective caps for central lines. Dr. Miller is Principal Investigator and serves as Vice Chair of Quality and Safety, Director of Division of Quality and Safety at the Johns Hopkins Children's Center. Dr. Miller had led and continues to lead efforts to transform the quality and safety of the delivery system at Johns Hopkins University and is a formally trained in Lean Six Sigma quality improvement as well as having her Masters of Science degree in clinical research. In addition, Dr. Aaron Milstone at Johns Hopkins University, director of pediatric hospital epidemiology and infection control and an accomplished researcher in pediatric infection prevention, will be a Co-Investigator on this proposal. Dr. Milstone led the recently published clinical trial work in Lancet describing the impact of chlorhexidine bathing on CLABSI and positive blood cultures in children in 10 PICUs. Dr. Elizabeth Colantuoni is a Biostatistician and Assistant Scientist in the Johns Hopkins Bloomberg School of Public Health.

The work will span four years. Year 1 Preparatory work will include establishing Institutional Review Board approval at each of the participating institutions, setting up data collection and submission processes, setting up distribution mechanisms for the intervention both to the clinics and then within each clinic to the homes, and educating providers, patients, and families on how to apply the CUROS® cap across all the participating institutions. Years 2, 3, and 4 will include two 12 month trial periods with a 3 month wash out period in between. The last 9 months of Year 4 will be used for data analysis and manuscript preparation.

Methods SPECIFIC AIM 1 and SPECIFIC AIM 2:

Specific Aim #1: Evaluate whether use of 70% isopropyl alcohol embedded protective caps on central lines reduces the rate of CLABSI in ambulatory pediatric hematology/oncology patients.

Hypothesis: Use of 70% isopropyl alcohol embedded protective caps on central lines will be associated with at least a 25% reduction in the ambulatory CLABSI rate for pediatric hematology/oncology patients.

Specific Aim #2: Evaluate whether use of 70% isopropyl alcohol embedded protective caps on central lines reduces the rate of all positive blood cultures in ambulatory pediatric hematology/oncology patients.

Hypothesis: Use of 70% isopropyl alcohol embedded protective caps on central lines will be associated with at least a 25% reduction in the positive blood culture rate at home for pediatric hematology/oncology patients.

Independent variables: The primary independent variable will be ambulatory CLABSI rates for Specific Aim #1 and all positive blood culture rates, defined as CLABSI rate + MBI-CLABSI rates + Secondary BSI rates + single positive blood culture (SPBC) rates, for Specific Aim #2. All of the participating units already devote Hospital Infection Control staff to identify and track all 3 of these types of ambulatory central line infections.

Dependent variable: The dependent variable for these Specific Aims will be the dichotomous assignment to either control or intervention arms where unit will receive both arms.

Data collection method: All Hematology/Oncology units will submit monthly aggregate clinic data on CLABSI, MBI-CLABSI, Secondary BSI and SPBC (numerators and denominators) via a web-based data entry tool.

Exploratory analyses: Events and line-days at the unit level will be calculated to summarize rates of infections (CLABSI and all infections) by treatment and period as well as by month to assess for any important trends. These trends will be evaluated using scatterplots and line plots, overall and separately by treatment arm and period. Summary statistics, such as mean, median, interquartile range and variance, for the monthly number of infection events and rates will be calculated for the overall sample and by treatment and period. In case missing data occurs in our analysis we will explore the relationship between missing data and the unit's observed data in months prior and our analysis methods will be valid under the assumptions that the missing data are generated completely at random or depend on the prior observed rates (missing at random). Our data integrity efforts and frequent contacts with this team will work to minimize any instances of missing data.

Multivariate analyses: Random effects Poisson regression models will be used to test for a treatment effect. Specifically, the monthly number of CLABSI (Specific Aim #1) or the monthly number of all infections (Specific Aim #2) will be modeled as a function of the dichotomous treatment assignment and an indicator for when the treatment arm was received (first or second 12 month period) with inclusion of an offset representing the monthly number of central line days and a random intercept for unit to account for the correlation of monthly rates of infections over time within the same unit. The models rely on two key assumptions: i) the infection rates follow a Poisson distribution where the mean rate is the same as the variance in the rate and ii) the correlation of the rates within a unit over time is exchangeable. These assumptions will be assessed via descriptive analyses and by adding a robust variance estimate clustering on the unit.

Methods, Specific Aim #3: To evaluate whether the use of 70% isopropyl alcohol embedded protective caps on central lines changes the distribution of bacteria isolated from blood cultures of ambulatory pediatric hematology/oncology patients.

Hypothesis: Use of 70% isopropyl alcohol embedded protective caps on central lines will be associated with altered microbial epidemiology for CLABSI, secondary blood steam infections, and single positive blood cultures at home for pediatric hematology/oncology patients.

Independent variables: Organisms isolated for all blood cultures (CLABSI + MBI-CLABSI + Secondary BSI + SPBC) in patients involved in this study will be collected from participating teams during both the Control and Intervention arms of the clinical trial and sorted into Gram Positive versus Gram Negative organisms.

Dependent variable: The dependent variable for this Specific Aim will be the dichotomous assignment to either control or intervention arms.

Data collection method: All Hematology/Oncology ambulatory care teams will submit the microbial pattern data for all positive blood cultures.

Analyses: The analysis would be a comparison of proportions of Gram positive organisms causing CLABSI, SPBC, and all positive blood cultures between the control and intervention study arms. Given that Gram positive organisms are the most common organisms causing CLABSI and SPBC in children, achieving a reduction in Gram positive organisms would be an important additional finding of this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* pediatric outpatients with either hematologic or oncologic diagnosis who have an external central line

Exclusion Criteria:

* none

Ages: 1 Day to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene R. Miller, MD, MSc, Principal Investigator — University Hospitals; Aaron Milstone, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (16):
- United States (16):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Colorado, Aurora, Colorado
  - Nemours Alfred Dupont Hospital for Children, Wilmington, Delaware
  - University of Florida Children's Hospital, Gainesville, Florida
  - Norton Children's Hospital, Louisville, Kentucky
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - St Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Montefiore, The Bronx, New York
  - Akron Children's Hospital, Akron, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Medical University of South Carolina Children's Hospital, Charleston, South Carolina
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Participating individuals are at the hospital level via hospital ambulatory central line infection rates

REFERENCES:
- [Derived] Milstone AM, Rosenberg C, Yenokyan G, Koontz DW, Miller MR; CCLIP Authorship Group. Alcohol-impregnated caps and ambulatory central-line-associated bloodstream infections (CLABSIs): A randomized clinical trial. Infect Control Hosp Epidemiol. 2021 Apr;42(4):431-439. doi: 10.1017/ice.2020.467. Epub 2020 Oct 12. PMID 33040755

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data was collected at the clinic level, there was no data collected at the participant level and therefore there are no participant numbers available for any results modules.
Units Other Than Participants: Clinics
Period: Intervention 1 (12 Months)
Arm/Group | Usual Care Only, Then Usual Care + 70% Isopropyl Alcohol | Usual Care + 70% Isopropyl Alcohol, Then Usual Care Only
Started | NA; 7 Clinics (Number of participants is not available for this study, only clinic-level data collected.) | NA; 9 Clinics (Number of participants is not available for this study, only clinic-level data collected.)
Completed | NA; 7 Clinics (Number of participants is not available for this study, only clinic-level data collected.) | NA; 9 Clinics (Number of participants is not available for this study, only clinic-level data collected.)
Not Completed | NA; 0 Clinics | NA; 0 Clinics
Period: Washout (2-3 Months)
Arm/Group | Usual Care Only, Then Usual Care + 70% Isopropyl Alcohol | Usual Care + 70% Isopropyl Alcohol, Then Usual Care Only
Started | NA; 7 Clinics (Number of participants is not available for this study, only clinic-level data collected.) | NA; 9 Clinics (Number of participants is not available for this study, only clinic-level data collected.)
Completed | NA; 7 Clinics (Number of participants is not available for this study, only clinic-level data collected.) | NA; 9 Clinics (Number of participants is not available for this study, only clinic-level data collected.)
Not Completed | NA; 0 Clinics | NA; 0 Clinics
Period: Intervention 2 (12 Months)
Arm/Group | Usual Care Only, Then Usual Care + 70% Isopropyl Alcohol | Usual Care + 70% Isopropyl Alcohol, Then Usual Care Only
Started | NA; 7 Clinics (Number of participants is not available for this study, only clinic-level data collected.) | NA; 9 Clinics (Number of participants is not available for this study, only clinic-level data collected.)
Completed | NA; 7 Clinics (Number of participants is not available for this study, only clinic-level data collected.) | NA; 9 Clinics (Number of participants is not available for this study, only clinic-level data collected.)
Not Completed | NA; 0 Clinics | NA; 0 Clinics

BASELINE CHARACTERISTICS:
Population: Number of participants is not available for this study, only clinic-level data collected.
Units Other Than Participants: Clinics
Groups:
- All Clinics: All 16 clinics included in this cluster-randomized trial.
Arm/Group | All Clinics
Number analyzed (Participants) | NA
Number analyzed (Clinics) | 16
Age, Customized [Median (Inter-Quartile Range); unit: percentage of participants] — Data collected and reported reflect the median percentage of participants across all clinics for each age category in the data table.
  percentage of participants
    < 2 years | 15 [10 to 19]
    2 - 5 years | 19 [15 to 22]
    6 - 11 years | 26 [24 to 29]
    ≥ 12 years | 41 [36 to 46]
Sex/Gender, Customized [Number; unit: percentage of participants]
  Female | 46
  Male | 54
Race (NIH/OMB) [Count of Units; unit: Clinics]
  American Indian or Alaska Native | NA — No race data was collected.
  Asian | NA — No race data was collected.
  Native Hawaiian or Other Pacific Islander | NA — No race data was collected.
  Black or African American | NA — No race data was collected.
  White | NA — No race data was collected.
  More than one race | NA — No race data was collected.
  Unknown or Not Reported | NA — No race data was collected.
Region of Enrollment [Number; unit: Clinics]
  United States | 16
Number of inpatient pediatric oncology beds [Median (Inter-Quartile Range); unit: beds] | 25 [20 to 34]
Number of annual pediatric oncology admissions [Median (Inter-Quartile Range); unit: admissions] | 1091 [727 to 1354]
Number of pediatric oncology ambulatory visits [Median (Inter-Quartile Range); unit: ambulatory visits] | 8552 [6790 to 11858]
Number of total inpatient days [Median (Inter-Quartile Range); unit: days] | 5640 [4664 to 8423]
Number of total Bone Marrow Transplant/Stem Cell [Median (Inter-Quartile Range); unit: transplants] | 32 [10 to 49]

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Central Line Associated Blood Stream Infections (CLABSI)
Description: To obtain rate of ambulatory central line associated blood stream infections in ambulatory patients
Time Frame: 2 years
Population: Number of participants is not available for this study, only clinic-level data collected.
Measure: Number; unit: infections
Units Other Than Participants: Clinics
Groups:
- Usual Care Only: Clinics using usual care only.
- Usual Care + 70% Isopropyl Alcohol: Clinics using usual care + 70% isopropyl alcohol.
Arm/Group | Usual Care Only | Usual Care + 70% Isopropyl Alcohol
Number analyzed (Participants) | NA | NA
Number analyzed (Clinics) | 16 | 16
infections
  Per Protocol | 113 | 84
  Intent-to-treat | 123 | 109

2. Secondary Outcome: Total Number of Mucosal Barrier Injury Central Line-associated Bloodstream Infections (MBI-CLABSI)
Description: To obtain rate of ambulatory Mucosal Barrier Injury central line-associated bloodstream infections (MBI-CLABSI)
Time Frame: 2 years
Population: Number of participants is not available for this study, only clinic-level data collected.
Measure: Number; unit: infections
Units Other Than Participants: Clinics
Arm/Group | Usual Care Only | Usual Care + 70% Isopropyl Alcohol
Number analyzed (Participants) | NA | NA
Number analyzed (Clinics) | 16 | 16
infections
  Per Protocol | 14 | 8
  Intent-to-treat | 16 | 10

3. Secondary Outcome: Total Number of Ambulatory Secondary Bloodstream Infections (Secondary BSI)
Description: To obtain rate of ambulatory secondary bloodstream infections
Time Frame: 2 years
Population: Number of participants is not available for this study, only clinic-level data collected.
Measure: Number; unit: secondary bloodstream infections
Units Other Than Participants: Clinics
Arm/Group | Usual Care Only | Usual Care + 70% Isopropyl Alcohol
Number analyzed (Participants) | NA | NA
Number analyzed (Clinics) | 16 | 16
secondary bloodstream infections
  Per Protocol | 11 | 0
  Intent-to-treat | 11 | 0

4. Secondary Outcome: Total Number of Ambulatory Single Positive Blood Cultures (SPBC)
Description: To obtain rate of ambulatory single positive blood culture (SPBC)
Time Frame: 2 years
Population: Number of participants is not available for this study, only clinic-level data collected.
Measure: Number; unit: single positive blood cultures
Units Other Than Participants: Clinics
Arm/Group | Usual Care Only | Usual Care + 70% Isopropyl Alcohol
Number analyzed (Participants) | NA | NA
Number analyzed (Clinics) | 16 | 16
single positive blood cultures
  Per Protocol | 29 | 42
  Intent-to-treat | 36 | 51

5. Secondary Outcome: Total Number of Ambulatory Positive Blood Culture
Description: To obtain rate of ambulatory positive blood culture rate
Time Frame: 2 years
Population: Number of participants is not available for this study, only clinic-level data collected.
Measure: Number; unit: positive blood cultures
Units Other Than Participants: Clinics
Arm/Group | Usual Care Only | Usual Care + 70% Isopropyl Alcohol
Number analyzed (Participants) | NA | NA
Number analyzed (Clinics) | 16 | 16
positive blood cultures
  Per Protocol | 167 | 134
  Intent-to-treat | 186 | 170

6. Secondary Outcome: Total Number of Acquired Pathogens
Description: Organism distribution of Gram positive bacteria, Gram negative bacteria, fungi, or other.
Time Frame: 2 years
Population: Number of participants is not available for this study, only clinic-level data collected.
Measure: Number; unit: microorganisms
Units Other Than Participants: Clinics
Arm/Group | Usual Care Only | Usual Care + 70% Isopropyl Alcohol
Number analyzed (Participants) | NA | NA
Number analyzed (Clinics) | 16 | 16
microorganisms
  Gram positive microorganisms | 69 | 63
  Gram negative microorganisms | 72 | 75
  Yeast | 3 | 1
  Mycobacterium | 2 | 1
  Other | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Clinics were asked to report any Adverse Events if they occurred and no Adverse Events were reported. The at Risk is entered as 0 because the precise number of participants from each clinic is unknown.
Arm/Group | All Clinics
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT02351258/Prot_SAP_000.pdf